CLINICAL TRIAL: NCT02451813
Title: The Relationship Between Needle Position and Injection Pressure During Femoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: StLukeNY
Record Dates: First submitted 2015-03-03; First posted 2015-05-22 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Orthopedic Disorders
Keywords: opening injection pressure; femoral nerve block; fascia iliaca; ultrasound guided nerve block
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): A 22 GA 5 cm nerve block needle will be advanced to the following conditions:
  1. Needle tip slightly indenting the fascia iliaca
  2. Needle tip advanced through fascia iliaca
  3. Needle tip slightly indenting the anterior surface of the femoral nerve
  4. Needle tip withdrawn 1 mm from nerve.
  At each of these conditions, 1 ml of dextrose solution will be injected and spread of injectate observed sonographically. A blinded observer will measure injection pressure. If opening pressure reaches 15 psi, this investigator will halt the injection. In addition, minimum threshold current required to elicit a motor response will be recorded for conditions 3 and 4.
  Interventions: Procedure: Apposition of needle bevel against femoral nerve

INTERVENTIONS:
Procedure: Apposition of needle bevel against femoral nerve — Indentation of femoral nerve and fascia iliaca by block needle and measurement of opening injection pressure during the controlled injection of 1 ml of dextrose (D5W) solution

SUMMARY:
Recent evidence suggests that injection pressure monitoring may be able to predict needle nerve contact in the brachial plexus nerve block model, but little is known about multifascicular nerves. The investigators hypothesize that injection pressure monitoring can reliably predict needle-nerve contact during femoral nerve block.

DETAILED DESCRIPTION:
Single center, observational study. Patients scheduled for elective lower limb surgery with femoral nerve block will be recruited. Femoral nerve will be identified using a linear ultrasound transducer. A 22 GA 5 cm nerve block needle will be inserted with bevel downward and advanced to the following conditions:

1. Needle tip slightly indenting the fascia iliaca lateral to the femoral nerve
2. Needle tip advanced through fascia iliaca
3. Needle tip slightly indenting the anterior surface of the femoral nerve
4. Needle tip withdrawn 1 mm from nerve.

At each of these conditions, 1 ml of dextrose solution will be injected via an automated pump at 10 ml/min and the spread of injectate observed sonographically. Simultaneously, a blinded observer will measure opening injection pressure using both an electronic and a mechanical transducer. If opening pressure reaches 15 psi, this investigator will halt the injection. In addition, minimum threshold current required to elicit a motor response will be recorded for conditions 3 and 4. Patients will be contacted at 7 days and asked about any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* ASA physical status I-III
* scheduled for lower limb surgery where femoral block is part of intended analgesic plan

Exclusion Criteria:

* Contraindication to femoral nerve block (e.g. infection)
* BMI > 35 kg/m2
* inability to communicate postoperative symptoms
* pre-existing neurologic deficits in the operative extremity
* allergy to local anesthetics
* history of opioid dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of high opening injection pressure (15 psi or greater) when needle tip in contact with nerve | 1 minute

SECONDARY OUTCOMES:
Incidence of high opening injection pressure (15 psi or greater) at other needle locations | 1 minute
Minimum threshold current to elicit a motor response with needle-nerve contact and needle disengagement | 1 minute
Incidence of paresthesias | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Malikah Latmore, MD, Study Director — Mount Sinai St. Luke's Mount Sinai Roosevelt Hospitals
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States